CLINICAL TRIAL: NCT00826436
Title: A Randomized, Placebo-Controlled, Double-Blind, Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of PRA-027 Administered Orally to Japanese Postmenopausal Women
Brief Title: Study Evaluating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PRA-027 in Japanese Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 3208A1-1008
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Uterine Leiomyomata (Fibroids)
MeSH Terms: conditions — Myofibroma; Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 8 subjects for Cohort 1
- 8 subjects for Cohort 2

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of ascending, multiple, oral doses of PRA-027 in Japanese postmenopausal women. The secondary purpose is to evaluate the PK and PD profile of multiple oral doses of PRA-027 in Japanese postmenopausal women.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Aged 35 to 65 years inclusive on study day 1 of the treatment period. Menopause may be spontaneous or due to surgery.

   Postmenopausal women are defined as follows:
   * Spontaneous amenorrhea must have begun by age 55 years.
   * Spontaneous amenorrhea must have initiated at least 6 months before study day 1 of the treatment period.
   * For subjects who have had spontaneous amenorrhea for at least 6 months but less than 12 months before screening, follicle-stimulating hormone (FSH) level must be ≥ 38 mIU/mL.
   * For subjects who have had spontaneous amenorrhea for 12 months or longer before screening, no FSH level determination is required.
   * For subjects who have had amenorrhea as a result of bilateral oophorectomy without hysterectomy; surgery must have occurred at least 6 months before screening. No FSH measurement is required. Subjects must provide evidence of the procedure by an operative report or by ultrasound scan. The date (month/year) of the subjects' last menstrual period must be determined and recorded on the source document.
2. Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and bodyweight ≥ 45 kg.

   BMI is calculated by taking the subject's weight, in kilograms, divided by the square of the subject's average height, in meters, at screening:BMI = weight (kg)/[Height (m)]2
3. Healthy, as determined by the investigator, on the basis of screening evaluations.
4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatinine levels should be below the upper limit of normal at screening.
5. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.
6. Have a high probability for compliance with and completion of the study.

EXCLUSION CRITERIA:

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Any significant cardiovascular, hepatic, renal, respiratory,gynecologic, gastrointestinal, endocrine, immunologic,dermatologic, hematologic, neurologic, or psychiatric disease.

   - Women with asymptomatic leiomyomata may be enrolled in the study.
3. Women who have undergone a hysterectomy.
4. Women with complex or simple ovarian cysts greater than 3 cm indiameter.
5. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article (eg, resection of liver, kidney, gallbladder, or gastrointestinal tract).
6. Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before receiving test article (treatment period study day 1).
7. History of drug abuse.
8. Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements.
9. History or presence of polycystic ovarian disease.
10. History of female infertility.
11. History or family history of arterial or venous thrombosis.
12. Any clinically significant deviation from normal limits in results of physical examinations, vital sign measurements, 12-lead electrocardiograms (ECGs), or clinical laboratory tests.
13. Demonstration of positive findings on orthostatic testing at screening. The definition of a positive finding is a ≥20 mm Hg decrease in systolic blood pressure, a ≥ 10 mm Hg decrease in diastolic blood pressure, or a ≥ 30 bpm increase in pulse, after standing for 3 minutes.
14. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
15. Positive findings from urine drug screening (eg, amphetamines,barbiturates, benzodiazepines, cannabinoids, cocaine, opiates and phencyclidine [PCP]).
16. History of any clinically important drug allergy or adverse drug reaction (eg, relapsing dermatitis, drug hypersensitivity, drug allergy, hypersensitivity to ingredient in the test articles, angioedemas)
17. Use of any investigational or prescription drug within 90 days before receiving test article (treatment period day 1)or prescription drug within 30 days before study day 1.
18. Consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or carbonated beverages) or alcoholic beverages within 48 hours before receiving test article (treatment period day 1).
19. Consumption of grapefruit or grapefruit-containing products within 72 hours before study day 1 (treatment period day 1).
20. Use of any over-the-counter drugs, including herbal supplements (except for the use of vitamins ≤ 100% of the recommended daily allowance), within 14 days before receiving test article (treatment period day 1).
21. Donation of blood within 90 days before study day 1.
22. Subjects deemed by the investigator to be inappropriate according for the inclusion in the study.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple oral doses of PRA-027 in postmenopausal women. | 28 days

SECONDARY OUTCOMES:
To evaluate the Pharmacokinetics and Pharmacodynamics profile of multiple oral doses of PRA-027 in postmenopausal women. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Kagoshima, Kagoshima-ken, Japan